CLINICAL TRIAL: NCT04775953
Title: Dalbavancin as an Option for Treatment of S. Aureus Bacteremia (DOTS): A Phase 2b, Multicenter, Randomized, Open-Label, Assessor-Blinded Superiority Study to Compare the Efficacy and Safety of Dalbavancin to Standard of Care Antibiotic Therapy for the Completion of Treatment of Patients With Complicated S. Aureus Bacteremia
Brief Title: DOTS: Dalbavancin as an Option for Treatment of Staphylococcus Aureus Bacteremia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0002; 5UM1AI104681-12 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2022-02-10

CONDITIONS: Staphylococcal Bacteraemia
Keywords: Bacteremia; Dalbavancin; DOTS; Efficacy; Safety; Staphylococcus aureus
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections | interventions — Cefazolin; dalbavancin; Daptomycin; Nafcillin; Oxacillin; Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Dalbavancin) (Experimental): Dalbavancin 1500 mg will be administrated intravenously (IV) over 30 (-/+10) minutes on Day 1 and 1500 mg IV over 30 (-/+10) minutes on Day 8, renally dose-adjusted to 1125 mg for subjects with Creatinine Clearance (CrCl) <30 and not on dialysis. N=100
  Interventions: Drug: Dalbavancin
- Arm 2 (Standard of Care) (Active Comparator): For Methicillin-sensitive Staphylococcus aureus (MSSA): nafcillin (2 g will be administrated intravenously (IV) every 4 hours for 4-6 weeks) OR oxacillin (2 g will be administrated intravenously (IV) every 4 hours for 4-6 weeks OR cefazolin (2 g will be administrated intravenously (IV) every 8 hours for 4-6 weeks) For Methicillin-resistant Staphylococcus aureus (MRSA): vancomycin (dose per local standard of care × 4-6 weeks) OR daptomycin (6-10 mg/kg will be administrated intravenously (IV) daily for 4-6 weeks). N=100
  Interventions: Drug: Cefazolin; Drug: Daptomycin; Drug: Nafcillin; Drug: Oxacillin; Drug: Vancomycin

INTERVENTIONS:
Drug: Cefazolin — Cefazolin is a semisynthetic cephalosporin analog with broad-spectrum antibiotic action due to inhibition of bacterial cell wall synthesis. Cefazolin (2 g will be administrated intravenously (IV) every 8 hours for 4-6 weeks)
  Arms: Arm 2 (Standard of Care)
Drug: Dalbavancin — A second-generation lipoglycopeptide antibiotic synthesized from a fermentation product of Nonomuraea species
  Arms: Arm 1 (Dalbavancin)
Drug: Daptomycin — Daptomycin (USA) or Cubicin (Spain) is a cyclic lipopeptide antibiotic that inhibits gram-positive bacteria. Daptomycin (6-10 mg/kg will be administrated intravenously (IV) daily for 4-6 weeks
  Arms: Arm 2 (Standard of Care)
Drug: Nafcillin — Nafcillin is a semi-synthetic antibiotic related to penicillin. Nafcillin (2 g will be administrated intravenously (IV) every 4 hours for 4-6 weeks)
  Arms: Arm 2 (Standard of Care)
Drug: Oxacillin — Oxacillin is an antibiotic used in resistant staphylococci infections. Oxacillin (2 g will be administrated intravenously (IV) every 4 hours for 4-6 weeks
  Arms: Arm 2 (Standard of Care)
Drug: Vancomycin — Vancomycin is a glycopeptide antibiotic product of the organism Amycolatopsis orientalis. Vancomycin (dose per local standard of care × 4-6 weeks)
  Arms: Arm 2 (Standard of Care)

SUMMARY:
This is a Phase 2b clinical study, multicenter, randomized, open-label, assessor-blinded, superiority study. The study will compare dalbavancin to standard of care antibiotic therapy for the completion of therapy in patients with complicated bacteremia or right-sided native valve Infective Endocarditis (IE) caused by S. aureus who have cleared their baseline bacteremia. Approximately 200 subjects will be randomized 1:1 to receive either dalbavancin or a standard of care antibiotic regimen that is based upon the identification and antibiotic susceptibility pattern of the baseline organism. Subjects randomized to the dalbavancin treatment group will receive 2 doses of dalbavancin intravenously (IV) 1 week apart (1500 mg on Day 1 and Day 8 after randomization, with renal dose adjustment if appropriate). Subjects randomized to the standard of care antibiotic therapy treatment group will receive an antibiotic regimen considered to be standard of care based on the methicillin susceptibility pattern of the pathogen isolated at baseline for a duration of 4 to 6 weeks and up to 8 weeks for patients with vertebral osteomyelitis/discitis. The primary objective is to compare the Desirability of Outcome Ranking (DOOR) at Day 70 of dalbavancin to that of standard of care antibiotic therapy used to consolidate therapy for the treatment of subjects with complicated S. aureus bacteremia in the intent-to-treat population (ITT).

DETAILED DESCRIPTION:
This is a Phase 2b clinical study, multicenter, randomized, open-label, assessor-blinded, superiority study. The study will compare dalbavancin to standard of care antibiotic therapy for the completion of therapy in patients with complicated bacteremia or right-sided native valve Infective Endocarditis (IE) caused by S. aureus who have cleared their baseline bacteremia. Approximately 200 subjects will be randomized 1:1 to receive either dalbavancin or a standard of care antibiotic regimen that is based upon the identification and antibiotic susceptibility pattern of the baseline organism. Subjects randomized to the dalbavancin treatment group will receive 2 doses of dalbavancin intravenously (IV) 1 week apart (1500 mg on Day 1 and Day 8 after randomization, with renal dose adjustment if appropriate). Subjects randomized to the standard of care antibiotic therapy treatment group will receive an antibiotic regimen considered to be standard of care based on the methicillin susceptibility pattern of the pathogen isolated at baseline for a duration of 4 to 6 weeks and up to 8 weeks for patients with vertebral osteomyelitis/discitis. The primary objective is to compare the Desirability of Outcome Ranking (DOOR) at Day 70 of dalbavancin to that of standard of care antibiotic therapy used to consolidate therapy for the treatment of subjects with complicated S. aureus bacteremia in the intent-to-treat population (ITT). The secondary objectives are 1) to compare the clinical outcomes of dalbavancin with the standard of care antibiotic therapy at day 70 in the modified intent-to-treat population (mITT). 2) to compare the safety of dalbavancin with that of the standard of care treatment in the modified intent-to-treat population (mITT). 3) to compare each individual component of the Desirability of Outcome Ranking (DOOR) outcome by treatment arm, in the intent-to-treat population.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient or legally authorized representative before the initiation of any study-specific procedures.
2. Patients > / = to 18 years old.
3. A diagnosis of complicated Staphylococcus aureus (either Methicillin-sensitive Staphylococcus aureus or Methicillin-resistant Staphylococcus aureus) bloodstream infection.
4. Treated with effective antibiotic therapy for at least 72 hours (maximum 10 days).*

   *Ten consecutive days prior to randomization is the maximum allowed treatment duration. If a subject has received intermittent or incomplete therapy earlier in the treatment course for this episode of S. aureus bacteremia, then discuss with the protocol PI and DMID Medical Officer prior to enrollment.
5. Subsequent defervescence for at least 24 hours and clearance of bacteremia from the qualifying pathogen (at Screening), with negative blood culture incubated for at least 48 hours.**

   **Two negative blood cultures incubated for 48 hours are preferred. However, if only a single blood culture set is drawn, no growth at 48 hours will be considered adequate to demonstrate clearance. If more than one culture set is drawn, all must show no growth at 48 hours to be considered evidence of clearance (e.g., 1 of 2 positive cultures would still be considered as ongoing bacteremia).
6. Provider willing to treat with either dalbavancin for two doses, or standard of care intravenous monotherapy for at least 4 and no more than 8 weeks from randomization.
7. Patients must be willing and able, if discharged, to return to the hospital or designated clinic for scheduled treatment, laboratory tests, or other procedures as required by the protocol.
8. According to the site Principal Investigator or sub-investigator assessment, patients must be expected to survive with appropriate antibiotic therapy and appropriate supportive care throughout the study.

Exclusion Criteria:

1. Uncomplicated bacteremia.*

   *Uncomplicated Staphylococcus aureus bacteremia is defined as all of the following: exclusion of endocarditis by echocardiography; catheter-associated bacteremia and removal of catheter; no implanted prostheses; follow-up blood cultures drawn within 48 hours after initial set that do not grow screening pathogen and all follow-up blood cultures thereafter do not grow the screening pathogen; defervescence within 72 hours of initiating effective therapy; and no evidence of metastatic sites of infection.
2. Infectious Central Nervous System events, including septic emboli, ischemic or hemorrhagic stroke, epidural abscess, or meningitis (prior/unrelated Central Nervous System events are not exclusion criteria).
3. Known or suspected left-sided endocarditis or presence of a perivalvular abscess.
4. Planned right-sided valve replacement surgery in the first 3 days following randomization.
5. Presence of prosthetic heart valve, cardiac device** UNLESS removal is planned within 4 days post-randomization.

   **Implantable cardioverter defibrillator (ICD), permanent pacemaker, valve support ring, ventricular assist device (VAD).
6. Presence of intravascular graft or intravascular material*** UNLESS removal is planned within 4 days post-randomization

   ***Excluding cardiac stents, inferior vena cava filters in place for >6 weeks, vascular stents in place for >6 weeks, non-hemodialysis grafts in place >90 days, and hemodialysis grafts not used within the past 12 months and not previously infected. A fistula constructed from native veins or a biologic vascular graft (without synthetic graft material) does not count as intravascular graft/material.
7. Infected prosthetic joint or extravascular hardware UNLESS removal is planned within 4 days post-randomization OR hardware was placed >60 days before bacteremia and clinically appears uninfected.
8. Polymicrobial bacteremia unless the non-Staphylococcus aureus organism is a contaminant.****

   ****Note: If a gram-negative bacteremia or fungemia develops after the qualifying S. aureus blood culture, AND the patient does not have right-sided endocarditis, AND the infection can be treated with an antibiotic without efficacy against the patient's S. aureus isolate (e.g. aztreonam), then the patient may remain eligible. Discussion with the DMID Medical Officer is strongly encouraged.
9. Significant hepatic insufficiency (Child-Pugh class C or aspartate transaminase (AST)/alanine aminotransferase (ALT) values >5x Upper Limit Normal at the time of randomization).
10. Immunosuppression*****

    *****On chemotherapy or immunotherapy for active hematologic malignancy expected to cause > 7 days of absolute neutrophil count (ANC) < 100 cells/mm3, recent bone marrow transplant (in the past 90 days), solid organ transplantation within prior 3 months or receipt of augmented immunosuppression for rejection within 3 months, chronic granulomatous disease, human immunodeficiency virus (HIV) infection with a cluster of differentiation 4 (CD4) cell count < 50 cells/mm3 based on last known measurement or patient-reported value.
11. History of hypersensitivity reaction to dalbavancin or other drugs of the glycopeptide class of antibiotics.
12. Treatment with either dalbavancin or oritavancin in the 60 days prior to enrollment.
13. Infection with Staphylococcus aureus not susceptible to dalbavancin (dalbavancin mean inhibitory concentration Minimum Inhibitory Concentration (MIC) > 0.25 µg/mL) or vancomycin (vancomycin Minimum Inhibitory Concentration (MIC) > 2 µg/mL).
14. Planned treatment with concomitant systemic antibacterial therapy with potential efficacy against the patient's qualifying Staphylococcus aureus isolate, other than that allowed in the protocol.
15. Pregnant/ nursing females.
16. Females of childbearing potential must have a negative pregnancy test****** within 48h of randomization and use effective contraception for trial duration.

    ******If the serum pregnancy test results cannot be obtained before randomization, a urine pregnancy test may be used for enrollment.
17. Other medical or psychiatric condition that may, in the judgment of the investigator, increase the risk of study participation or interfere with interpretation of study results.
18. Unwilling or unable to follow study procedures.
19. Treatment with an investigational drug within 30 days preceding the first dose of study medication.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (23):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - University of California Davis Medical Center - Internal Medicine - Infectious Disease, Sacramento, California
  - Harbor UCLA Medical Center - Medicine - Infectious Diseases, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - University of Florida Health - Shands Hospital - Division of Infectious Diseases and Global Medicine, Gainesville, Florida
  - University of South Florida Health - Internal Medicine, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Health - Ochsner Medical Center - Department of Infectious Diseases, New Orleans, Louisiana
  - Henry Ford Health System - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health - Infectious Disease, Royal Oak, Michigan
  - University of Nebraska Medical Center - Infectious Diseases, Omaha, Nebraska
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - New York Presbyterian Hospital - Weill Cornell Medical Center - Infectious Diseases, New York, New York
  - SUNY Upstate Medical University - Infectious Disease Division, Syracuse, New York
  - Atrium Health ID Consultants & Infusion Care Specialists, Charlotte, North Carolina
  - Duke University Hospital - Infectious Diseases, Durham, North Carolina
  - East Carolina University - Infectious Diseases and Tropical/Travel Medicine Clinic, Greenville, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health and Science University - Adult Infectious Diseases Clinic, Portland, Oregon
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - Prisma Health - Greenville Health System - Infectious Disease, Greenville, South Carolina
  - The University of Texas - MD Anderson Cancer Center - Infectious Diseases, Houston, Texas
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
- McGill University Health Centre, Montreal, Canada

REFERENCES:
- [Derived] Turner NA, Hamasaki T, Doernberg SB, Lodise TP, King HA, Ghazaryan V, Cosgrove SE, Jenkins TC, Liu C, Sharma S, Zaharoff S, Wahid L, Renard VJ, Cook P, Raad I, Hachem R, Chaftari AM, Sims M, DeMarco C, Miller LG, McCarthy MW, Morse CG, Lucasti C, Forrest GN, Cherabuddi K, Polk C, Fazili T, Rupp ME, Thompson GR 3rd, Kim K, Strnad L, Schnee AE, McKinnell JA, Ramesh M, Silveira FP, McCarty TP, Lee TC, McDonald EG, Paolino K, Wiegand K, Wall A, Riccobene T, Patel R, Rappo U, Evans S, Chambers HF, Fowler VG Jr, Holland TL; Antibacterial Resistance Leadership Group. Dalbavancin for Treatment of Staphylococcus aureus Bacteremia: The DOTS Randomized Clinical Trial. JAMA. 2025 Aug 13:e2512543. doi: 10.1001/jama.2025.12543. Online ahead of print. PMID 40802264
- [Derived] Turner NA, Zaharoff S, King H, Evans S, Hamasaki T, Lodise T, Ghazaryan V, Beresnev T, Riccobene T, Patel R, Doernberg SB, Rappo U, Fowler VG Jr, Holland TL; Antibacterial Resistance Leadership Group (ARLG). Dalbavancin as an option for treatment of S. aureus bacteremia (DOTS): study protocol for a phase 2b, multicenter, randomized, open-label clinical trial. Trials. 2022 May 16;23(1):407. doi: 10.1186/s13063-022-06370-1. PMID 35578360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 23 clinical sites within the United States and Canada. The first participant was enrolled on April 22, 2021, and the last participant was enrolled on July 6, 2023.
Groups:
- Dalbavancin: Dalbavancin 1500 mg administrated intravenously (IV) over 30 (-/+10) minutes on Day 1 and 1500 mg IV over 30 (-/+10) minutes on Day 8, renally dose-adjusted to 1125 mg for participants with Creatinine Clearance (CrCl) <30 and not on dialysis.
  Dalbavancin: A second-generation lipoglycopeptide antibiotic synthesized from a fermentation product of Nonomuraea species
- Standard of Care: For Methicillin-sensitive Staphylococcus aureus (MSSA): nafcillin (2 g administrated intravenously (IV) every 4 hours for 4-6 weeks) OR oxacillin (2 g administrated IV every 4 hours for 4-6 weeks OR cefazolin (2 g administrated IV every 8 hours for 4-6 weeks).
  For Methicillin-resistant Staphylococcus aureus (MRSA): vancomycin (dose per local standard of care × 4-6 weeks) OR daptomycin (6-10 mg/kg administrated IV daily for 4-6 weeks).
  Cefazolin: Cefazolin is a semisynthetic cephalosporin analog with broad-spectrum antibiotic action due to inhibition of bacterial cell wall synthesis.
  Daptomycin: Daptomycin (USA) or Cubicin (Spain) is a cyclic lipopeptide antibiotic that inhibits gram-positive bacteria.
  Nafcillin: Nafcillin is a semi-synthetic antibiotic related to penicillin.
  Oxacillin: Oxacillin is an antibiotic used in resistant staphylococci infections.
  Vancomycin: Vancomycin is a glycopeptide antibiotic product of the organism Amycolatopsis orientalis.
Period: Overall Study
Arm/Group | Dalbavancin | Standard of Care
Started | 100 | 100
Completed | 84 | 81
Not Completed | 16 | 19
Not completed — Lost to Follow-up | 6 | 11
Not completed — Death | 5 | 4
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Participant non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin | Standard of Care | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (15.7) | 54.0 (16.8) | 54.1 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 70 | 68 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 84 | 84 | 168
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 29 | 49
  White | 68 | 69 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 0 | 2
  United States | 98 | 100 | 198
Baseline Pathogen [Count of Participants; unit: Participants]
  MRSA | 34 | 32 | 66
  MSSA | 66 | 68 | 134
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.83 (6.91) | 29.03 (8.08) | 28.93 (7.50)

OUTCOME MEASURES:

1. Primary Outcome: Desirability of Outcome Ranking (DOOR)
Description: DOOR is a composite endpoint assessed by: (1) Clinical Failure: Lack of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated for its treatment; (2) Infectious Complications such as: Endocarditis, New evidence of metastatic foci of infection, relapse - isolation of baseline S. aureus pathogen from a blood culture drawn after randomization, readmission for subsequent care of indication under study, need for additional unplanned source control procedures, or change in antibiotic therapy due to inadequate clinical response; (3) Serious Adverse Events (SAEs); (4) Adverse Events (AEs) Leading to Study Drug Discontinuation; and (5) Death. Clinical failure and infectious complications were assessed by a blinded adjudication committee. Participants missing clinical failure were treated as having clinical failure for calculation of DOOR.
Time Frame: Day 70
Population: The intent-to-treat (ITT) population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants
  Rank 1: Alive with none of clinical failure, infectious comp, or SAE or AE leading to trt discont | 49 | 49
  Rank 2: Alive with one of clinical failure, infectious comp, or SAE or AE leading to trt discont | 34 | 37
  Rank 3: Alive with two of clinical failure, infectious comp, or SAE or AE leading to trt discont | 9 | 7
  Rank 4: Alive with all of clinical failure, infectious comp, and SAE or AE leading to trt discont | 4 | 3
  Rank 5: Death | 4 | 4
Statistical Analysis 1: Comparison: Dalbavancin vs Standard of Care; Null Hypothesis: Probability that a participant in the dalbavancin arm has a better DOOR than a participant in the standard of care arm plus one-half the probability of equal DOOR is 50% (i.e., no difference in DOOR); Test type: Superiority — For participants with the same DOOR, quality-of-life (QoL) was used as a tiebreaker and was calculated as change from baseline QoL to Day 70 QoL score, as assessed by questions from the PROMIS physical function item bank (PROMIS Item Bank v2.0, short form 6b) on the Antibacterial Resistance Leadership Group (ARLG) Bloodstream Infection QoL Measure. Superiority of dalbavancin is concluded if the lower bound of the 95% confidence interval for the DOOR probability is greater than 50%; Pr(Better DOOR in dalbavancin arm) = 47.70, 95% CI 2-sided [39.84 to 55.68] — The DOOR probability is calculated using the Wilcoxon-Mann-Whitney statistic corrected for ties

2. Secondary Outcome: Frequency of Clinical Efficacy
Description: Number of participants that had clinical efficacy at Day 70. Clinical efficacy is defined as none of: (1) Clinical Failure: Lack of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated for its treatment; (2) Infectious Complications such as: Endocarditis, New evidence of metastatic foci of infection, relapse - isolation of baseline S. aureus pathogen from a blood culture drawn after randomization, readmission for subsequent care of indication under study, need for additional unplanned source control procedures, or change in antibiotic therapy due to inadequate clinical response; and (3) Death. Clinical failure and infectious complications are assessed by a blinded adjudication committee. Participants missing clinical failure are treated as not having clinical efficacy.
Time Frame: Day 70
Population: The modified intent-to-treat (mITT) population includes all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 73 | 72
Statistical Analysis 1: Comparison: Dalbavancin vs Standard of Care; Null Hypothesis: The proportion of clinical efficacy in the dalbavancin arm minus the proportion of clinical efficacy in the standard of care arm is -20%; Test type: Non-Inferiority — The non-inferiority margin is -20%. Non-inferiority of dalbavancin is concluded if the lower limit of the 95% confidence interval for the difference in proportions of clinical efficacy is greater than -20%; Risk Difference (RD) = 1, 95% CI 2-sided [-12 to 14] — Difference in proportions of clinical efficacy for dalbavancin compared to standard of care and 95% confidence interval obtained from a linear regression model

3. Secondary Outcome: Frequency of SAEs
Description: Number of participants that experience any SAEs from Day 1 to study completion (Day 70 or Day 180 for participants in the osteomyelitis subset). An AE is considered serious if, in the view of either the site principal investigator or sponsor, it results in: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 180
Population: The mITT population includes all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 43 | 37

4. Secondary Outcome: Frequency of AEs Leading to Study Drug Discontinuation
Description: Number of participants that experience any AEs leading to study drug discontinuation from Day 1 to study completion (Day 70 or Day 180 for participants in the osteomyelitis subset).
Time Frame: Day 1 through Day 180
Population: The mITT population includes all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 3 | 12

5. Secondary Outcome: Frequency of Clinical Failure (A Component of DOOR)
Description: Number of participants who had clinical failure at Day 70, used for DOOR at Day 70. Clinical Failure is defined as lack of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated for its treatment. Clinical failure is assessed by a blinded adjudication committee. Participants missing clinical failure are treated as having clinical failure.
Time Frame: Day 70
Population: The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 20 | 22

6. Secondary Outcome: Frequency of Infectious Complications (A Component of DOOR)
Description: Number of participants that experience any infectious complications from Day 1 through Day 70, used for DOOR at Day 70. Infectious complications include endocarditis, new evidence of metastatic foci of infection, relapse - isolation of baseline S. aureus pathogen from a blood culture drawn after randomization, readmission for subsequent care of indication under study, need for additional unplanned source control procedures, or change in antibiotic therapy due to inadequate clinical response. Infectious complications are assessed by a blinded adjudication committee.
Time Frame: Day 1 through Day 70
Population: The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 13 | 12

7. Secondary Outcome: Frequency of SAEs (A Component of DOOR)
Description: Number of participants that experience any SAEs from Day 1 to Day 70, used for DOOR at Day 70. An AE is considered serious if, in the view of either the site principal investigator or sponsor, it results in: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 70
Population: The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 40 | 34

8. Secondary Outcome: Frequency of AEs Leading to Study Drug Discontinuation (A Component of DOOR)
Description: Number of participants that experience any AEs leading to study drug discontinuation from Day 1 to Day 70, used for DOOR at Day 70.
Time Frame: Day 1 through Day 70
Population: The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 3 | 12

9. Secondary Outcome: Frequency of All-Cause Mortality (A Component of DOOR)
Description: Number of participants who passed away from Day 1 to Day 70, used for DOOR at Day 70.
Time Frame: Day 1 through Day 70
Population: The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: All unsolicited AEs grade 3 or higher, including laboratory abnormalities, as well as adverse events of special interest (AESIs) of any severity from time of first dose of study drug (i.e., dalbavancin or standard of care antibiotic) after randomization through follow-up (Day 70 or Day 180 for participants in osteomyelitis subset) were reported.
Arm/Group | Dalbavancin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 5/100 | 4/100
Serious Adverse Events (participants affected / at risk) | 43/100 | 37/100
Other Adverse Events (participants affected / at risk) | 5/100 | 1/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalbavancin (N=100) | Standard of Care (N=100)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (3) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (2) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Diabetic foot infection (Infections and infestations) | 2 (2) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 5 (5)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 1 (3) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0)
Proteus infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Septic pulmonary embolism (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Splenic abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 4 (4)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalbavancin (N=100) | Standard of Care (N=100)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT04775953/Prot_001.pdf
  • Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT04775953/SAP_002.pdf
  • Informed Consent Form (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT04775953/ICF_000.pdf